CLINICAL TRIAL: NCT02320968
Title: Sleep Position Reduces Acid Reflux and Decreases Extraesophageal Reflux Symptoms: A Non-randomized Prospective Study of the Amenity Health MedclineTM Sleep Assist Device
Brief Title: Sleep Position May Reduce Acid Reflux Symptoms at Night
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: low recruitment
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: Amenity Health, Inc. (Industry)
Responsible Party: Principal Investigator, Michael Vaezi, Principal Investigator, Vanderbilt University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 141619
Record Dates: First submitted 2014-12-11; First posted 2014-12-19 (Estimated); Last update posted 2017-05-01 (Actual); Status verified 2017-04

CONDITIONS: Extra-esophageal Reflux

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with nocturnal extraesophageal reflux (Experimental): This is a non-randomized study to evaluate the effectiveness of the MedclineTM Sleep Assist Device on patients who experience nocturnal extraesophageal reflux. All patients will receive the device. Participants will serve as their own controls while undergoing 96-hour pH monitoring. Participants will follow their regular sleep position patterns on Days 1 and 2 of the study and will use the sleep assist device on Days 3 and 4. pH data and patient report of symptoms will be evaluated during the initial 96 hours of the study to capture physiologic results. All participants will use the sleep assist device for the remainder of the study to determine if a reduction in overall reflux symptom index (RSI) is achieved.
  Interventions: Other: MedclineTM Sleep Assist Pillow

INTERVENTIONS:
Other: MedclineTM Sleep Assist Pillow — The pillow is designed so that the sleeper can have proper upper-body elevation while sleeping on his or her left side without the need for placing blocks under the head of the bed and bothering anyone else who may be sleeping in the bed. The pillow supports the patient's head, back and body to provide comfort while reducing or relieving acid reflux symptoms during sleep.

SUMMARY:
This study is designed to determine if the addition of the MedclineTM Sleep Assist Device will decrease night-time gastroesophageal reflux disease events.

DETAILED DESCRIPTION:
The MedcineTM Sleep Assist Device was recently developed by Amenity Health, Inc and is designed to elevate the head and torso and maintain a patient in the left-lateral position in order to decrease night-time/nocturnal acid reflux. The MedcineTM Sleep Assist Device is composed of a 9-inch incline base and a wrap-around body pillow. Traditionally wedge pillows have been recommended for patients with acid reflux. The addition of the body pillow helps to maintain the patient in the left-lateral position (LLP) during sleep, which has been shown to reduce night-time reflux compared to wedge alone, right lateral position and/or sleeping flat.

In healthy controls, sleeping in the left-lateral position with this device system significantly decreased esophageal acid exposure and overall episodes of acid reflux. To date, there has been no study in patients with extra-esophageal reflux (EER) and nocturnal heartburn.

Primary Objectives The primary objective of the this study is to evaluate the effect of a reflux pillow on esophageal acid exposure in patients complaining of nocturnal EER.

Secondary Objectives To evaluate the effect of the reflux pillow on nocturnal EER symptoms, sleep quality, daytime EER symptoms, and overall quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients between the ages of 18 and 65;
* Between 5'4" and 6'2"
* Body Mass Index<32
* Willing and able to provide written informed consent;
* Understands the clinical study requirements and is able to comply with the follow-up schedule set forth in the protocol;
* Clinically diagnosed with gastroesophageal reflux disease with extra-esophageal symptoms (i.e. chronic cough, choking, aspiration, chronic post nasal drip, globus, sore throat, throat clearing);
* Presents with Reflux Symptom Index (RSI) > 13;
* Undergoing Esophagogastroduodenoscopy (EGD) as part of routine care;
* Undergoing 96-hour pH monitoring via BRAVO capsule as part of routine care.

Exclusion Criteria:

* Currently being treated with another investigational medical device and/or drug;
* Currently receiving treatment for sleep apnea with continuous positive airway pressure (CPAP);
* Female patients who are of child-bearing potential and not using an acceptable method of birth control, or is pregnant or breast-feeding;
* Suspected esophageal cancer;
* Confirmed nasopharyngeal cancer;
* Previously undergone Nissen Fundoplication;
* Hiatal hernia > 4 cm

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-12; Primary Completion 2017-03-01 (Actual); Study Completion 2017-03-01 (Actual)

PRIMARY OUTCOMES:
Number of patients with reduced esophageal acid exposure during sleep | 30 days
  The patient will use the sleep assist device from days 3 - 30 and will complete various questionnaires at weeks 2 and 4 to determine if night-time reflux symptoms were improved.

SECONDARY OUTCOMES:
Number of patients with improved sleep quality | 30 days
  The patient will use the sleep assist device from days 3 - 30 and will complete various questionnaires at weeks 2 and 4 to determine if sleep quality and overall quality of life was improved.
Number of patients with improved daytime extraesphageal reflux symptoms | 30 days
  The patient will use the sleep assist device from days 3 - 30 and will complete various questionnaires at weeks 2 and 4 to determine if sleep quality and overall quality of life was improved.

CONTACTS AND LOCATIONS:
Overall Officials: Michael F Vaezi, MD,PhD, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University Medical Center, Endoscopy Lab, TVC 1410, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No